CLINICAL TRIAL: NCT02724176
Title: Potential Role for Carbon Nanoparticles to Guide Central Neck Dissection in Patients With Papillary Thyroid Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Wenbin Yu, department of head neck, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BJ20161206
Record Dates: First submitted 2016-03-18; First posted 2016-03-31 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- carbon nanoparticles (Experimental): 0.1 ml of CN suspension was injected per spot into the tissue surrounding the tumor using a skin test syringe. Two or three randomly selected spots were injected slowly for each tumor, and the total amount injected was no more than 0.5 mL per lobe.
  Interventions: Drug: carbon nanoparticles

INTERVENTIONS:
Drug: carbon nanoparticles — 0.1 ml of CN suspension was injected per spot into the tissue surrounding the tumor using a skin test syringe. Two or three randomly selected spots were injected slowly for each tumor, and the total amount injected was no more than 0.5 mL per lobe.
  Other Names: normal saline

SUMMARY:
Papillary thyroid cancer (PTC) is the most common subtype of thyroid cancer.

The most common site of PTC nodal metastases is the central neck, which has a reported rate of lymph node metastases as high as 50%~70%.

Central neck dissection has important value to ensure accurate clinical staging and surgical planning.

As a novel lymphatic tracer, carbon nanoparticles (CN) have been applied successfully in the detection of sentinel lymph nodes in breast and gastric cancers, while not been used as a lymphatic tracer for PTC. The goal of this study was to evaluate whether the use of CN facilitates the detection of lymph nodes, increases the number of metastatic lymph nodes removed, accurately reflects the metastatic condition of the central neck, and has the potential to protect the parathyroid glands.

DETAILED DESCRIPTION:
Thyroid cancer is the most common endocrine malignancy. It is estimated that 96% of all new endocrine organ cancers will originate from the thyroid gland, resulting in approximately 63,000 new cases in 2014 in the US1. Among them, papillary thyroid cancer (PTC) is the most common subtype of thyroid cancer, accounting for more than 90% of all thyroid cancers. The incidence of PTC has been increasing in recent years, largely because of advances in early detection with ultrasonography and fine-needle aspiration biopsy1-4. The most effective treatment for PTC is the complete removal of the primary tumor and the metastatic regional lymph nodes, which is a prerequisite for other adjuvant therapies. Cervical lymph node metastases are quite common in PTC and have been reported to occur in 12-81% of patients with PTC5. The most common site of PTC nodal metastases is the central neck, which has a reported rate of lymph node metastases as high as 50%~70%5. Lymph node metastases in this area are difficult to identify preoperatively because the lymph nodes typically do not appear abnormal on preoperative imaging6,7.

Routine dissection of the central neck compartment is still controversial due to uncertain prognostic value of preserving clinically non-apparent lymph node metastasis1,8, central neck dissection has important value to ensure accurate clinical staging and surgical planning. According to previously published data, prophylactic central dissection has been suggested to improve disease-specific survival and to decrease local recurrence9,10 as well as post-treatment thyroglobulin levels9,11. Neck dissection also informs postoperative treatment, follow-up programs, assessment of recurrence risk, and prognosis12. However, routine neck dissection is controversial because of the uncertain effect on prognosis of clinically non-apparent lymph node metastases and because of complications, such as damage to the parathyroid glands, hypoparathyroidism, temporary/permanent recurrent laryngeal nerve injury, and tracheal or esophageal injury, that may profoundly influence a patient's qual¬ity of life.

Methylene blue has been used in the detection of sentinel lymph nodes in thyroid cancer, but methylene blue can also stain parathyroid glands, thyroid tissue, and fat, which can make the anatomic boundaries unclear and thereby restrict the use of methylene blue in PTC. As a novel lymphatic tracer13,14, carbon nanoparticles (CN) have been applied successfully in the detection of sentinel lymph nodes in breast and gastric cancers, while not been used as a lymphatic tracer for PTC. Thus, investigators hypothesized that CN may have clinical value in thyroid cancer as a novel lymph node tracer to guide central neck dissection. The goal of this study was to evaluate whether the use of CN facilitates the detection of lymph nodes, increases the number of metastatic lymph nodes removed, accurately reflects the metastatic condition of the central neck, and has the potential to protect the parathyroid glands. In this study, investigators evaluated the clinical value of CN in acquiring a more accurate reflection of the central neck lymph node status and in guiding central neck dissection.

ELIGIBILITY:
Inclusion Criteria:

* All patients were diagnosed with PTC by preoperative fine needle aspiration cytology,
* Underwent the initial operation in our department, and had all tumors located in one lobe.
* PTC with a tumor between 1 and 4 cm

Exclusion Criteria:

* Nonthyroid cancer,
* Previous thyroid or parathyroid surgery
* Preoperative hypoparathyroidism or hypocalcemia
* Pregnancy or lactation
* Presence or suspicion of lateral neck lymph node metastasis,
* Age under 18 years
* Noncompliance with the follow-up protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2012-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
lymph node metastatic rates between the carbon nanoparticles and control group | one year
total dissected lymph nodes less than 5mm between the carbon nanoparticles and control group | one year
the number of metastatic lymph nodes with diameter < 5mm between the carbon nanoparticles and control group | one year

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Yu, MD, Study Chair — Department of head neck

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang K, Luo D, Huang M, Long M, Peng X, Li H. Protection of parathyroid function using carbon nanoparticles during thyroid surgery. Otolaryngol Head Neck Surg. 2013 Dec;149(6):845-50. doi: 10.1177/0194599813509779. Epub 2013 Oct 25. PMID 24163324
- [Result] Hao RT, Chen J, Zhao LH, Liu C, Wang OC, Huang GL, Zhang XH, Zhao J. Sentinel lymph node biopsy using carbon nanoparticles for Chinese patients with papillary thyroid microcarcinoma. Eur J Surg Oncol. 2012 Aug;38(8):718-24. doi: 10.1016/j.ejso.2012.02.001. Epub 2012 Apr 20. PMID 22521260
- [Result] Cai HK, He HF, Tian W, Zhou MQ, Hu Y, Deng YC. Colorectal cancer lymph node staining by activated carbon nanoparticles suspension in vivo or methylene blue in vitro. World J Gastroenterol. 2012 Nov 14;18(42):6148-54. doi: 10.3748/wjg.v18.i42.6148. PMID 23155345